CLINICAL TRIAL: NCT00077844
Title: An International Phase 2-3, Stratified, Randomized, Open-label, Parallel-group Clinical Trial to Evaluate the Safety and Efficacy of a Single Intravenous Bolus of Enoxaparin Versus Intravenous Unfractionated Heparin in Patients Undergoing Non-emergent Percutaneous Coronary Intervention
Brief Title: Safety and Efficacy of Enoxaparin in Percutaneous Coronary Intervention (PCI) Patients, an International Randomized Evaluation (STEEPLE)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XRP4563_4001; EudraCT #: 2004-003743-44
Record Dates: First submitted 2004-02-12; First posted 2004-02-18 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Percutaneous Coronary Intervention
MeSH Terms: interventions — enoxaparin sodium

INTERVENTIONS:
Drug: Enoxaparin sodium

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intravenous enoxaparin versus intravenous unfractionated heparin (UFH) in patients undergoing non-emergent PCI, as assessed by measuring the incidence of non-coronary artery bypass graft (CABG) major and minor bleeding.

ELIGIBILITY:
INCLUSION CRITERIA

* Male or non-pregnant female greater than or equal to 18 years of age
* Undergoing non-emergent single or multiple sites/vessels PCI during the same procedure
* PCI to be performed with a femoral approach

EXCLUSION CRITERIA

* Known or suspected pregnancy in women of childbearing potential
* Thrombolytic therapy within the previous 24 hours
* Undergoing primary PCI for ongoing ST-segment elevation myocardial infarction (STEMI)
* Undergoing rescue PCI after failed thrombolysis
* Any other elective PCI scheduled within the following 30 days after the index PCI
* Increased bleeding risk: ischemic stroke within the last year or any previous hemorrhagic stroke, intracranial tumor or aneurysm; recent (<1 month) trauma or major surgery (including bypass surgery); active bleeding
* Uncontrolled arterial hypertension
* Recent (<48 hours) or planned spinal/epidural anesthesia or puncture
* Impaired haemostasis: known International Normalized Ratio (INR) >1.5; past or present bleeding disorder (including congenital bleeding disorders such as von Willebrand's disease or hemophilia, acquired bleeding disorders, and unexplained clinically significant bleeding disorders), thrombocytopenia (platelet count <100,000/µL)
* History of hypersensitivity or contraindication to heparin or LMWH
* Treatment with oral anticoagulant therapy within 72 hours prior to inclusion or current need for vitamin-K antagonist therapy
* Treatment with a direct thrombin inhibitor, low molecular weight heparin, or unfractionated heparin within the 24 hours preceding enrolment
* Use of abciximab within the previous 7 days or, tirofiban, or eptifibatide within the past 12 hours of index PCI
* Inability to give informed consent or high likelihood of being unavailable for follow-up
* Treatment with other investigational agents or devices within the previous 30 days, planned use of investigational drugs or devices, or previous enrollment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3532 (Estimated)
Dates: Start 2004-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
the composite of non-CABG major and minor bleeding | up to H48 after index PCI

SECONDARY OUTCOMES:
success rate of achieving ACT target range | at the beginning and end of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Luc Sagnard, Study Director — Sanofi

REFERENCES:
- [Result] Montalescot G, White HD, Gallo R, Cohen M, Steg PG, Aylward PE, Bode C, Chiariello M, King SB 3rd, Harrington RA, Desmet WJ, Macaya C, Steinhubl SR; STEEPLE Investigators. Enoxaparin versus unfractionated heparin in elective percutaneous coronary intervention. N Engl J Med. 2006 Sep 7;355(10):1006-17. doi: 10.1056/NEJMoa052711. PMID 16957147
- [Result] Montalescot G, Cohen M, Salette G, Desmet WJ, Macaya C, Aylward PE, Steg PG, White HD, Gallo R, Steinhubl SR; STEEPLE Investigators. Impact of anticoagulation levels on outcomes in patients undergoing elective percutaneous coronary intervention: insights from the STEEPLE trial. Eur Heart J. 2008 Feb;29(4):462-71. doi: 10.1093/eurheartj/ehn008. PMID 18276619
- [Derived] White HD, Aylward PE, Gallo R, Bode C, Steg G, Steinhubl SR, Montalescot G; STEEPLE Investigators. Hematomas of at least 5 cm and outcomes in patients undergoing elective percutaneous coronary intervention: insights from the SafeTy and Efficacy of Enoxaparin in PCI patients, an internationaL randomized Evaluation (STEEPLE) trial. Am Heart J. 2010 Jan;159(1):110-6. doi: 10.1016/j.ahj.2009.10.034. PMID 20102875
- [Derived] Montalescot G, Gallo R, White HD, Cohen M, Steg PG, Aylward PE, Bode C, Chiariello M, King SB 3rd, Harrington RA, Desmet WJ, Macaya C, Steinhubl SR; STEEPLE Investigators. Enoxaparin versus unfractionated heparin in elective percutaneous coronary intervention 1-year results from the STEEPLE (SafeTy and efficacy of enoxaparin in percutaneous coronary intervention patients, an international randomized evaluation) trial. JACC Cardiovasc Interv. 2009 Nov;2(11):1083-91. doi: 10.1016/j.jcin.2009.08.016. PMID 19926048
- [Derived] White HD, Gallo R, Cohen M, Steg PG, Aylward PE, Bode C, Steinhubl S, Montalescot G. The use of intravenous enoxaparin in elective percutaneous coronary intervention in patients with renal impairment: results from the SafeTy and Efficacy of Enoxaparin in PCI patients, an internationaL randomized Evaluation (STEEPLE) trial. Am Heart J. 2009 Jan;157(1):125-31. doi: 10.1016/j.ahj.2008.08.019. Epub 2008 Nov 12. PMID 19081408